CLINICAL TRIAL: NCT00570362
Title: Evaluation of Systemic Glutathione Level in Patients With Normal Tension Glaucoma
Brief Title: Systemic Glutathione Level in Normal Tension Glaucoma
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Jung-Il Moon, St.Mary's Hospital, College of Medicine, The Catholic University of Korea
Other Study IDs: Merck-001; CMCEYE-GSH
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2007-12

CONDITIONS: Normal Tension Glaucoma
Keywords: Normal tension glaucoma; Glutathione; Antioxidant
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether systemic glutathione level is decreased in patients with normal tension glaucoma.

DETAILED DESCRIPTION:
Normal tension glaucoma is one of the most common cause of primary open angle glaucoma in Korea. Even though, we still do not know what the cause is. Only IOP-lowering drugs are the currently available therapeutic method. Glutathione is one of the mostly high concentrated intracellular antioxidants. We find apoptosis of neuronal cell in the mouse retina by systemic depletion of glutathione using buthionine sulfoximine. Glutathione is also known to be reduced in primary open angle glaucoma with high IOP. So we are planning to evaluate systemic glutathione level in normal tension glaucoma.

Blood samples will be obtained by venipuncture to the antecubital vein of normal tension glaucoma patients and age-matched normal controls. Five milliliters of blood will be collected in EDTA-treated tubes (to prevent oxidation). Thirty microliters of blood will be then transferred into centrifuge tubes, and will be added 33.3 microliter of 5-sulfosalicylic acid (SSA), 100mg/mL within 10 minutes from the blood collection.Each sample will be then diluted with 936.7 microliter sodium phosphate buffer (pH 7.5), and the content of each tube will be mixed rapidly in a centrifuge at 13,000 rpm for 5 minutes. A portion of supernatant (150 microliter) will be then collected into clean centrifuge tubes and immediately cooled at -70°C. To each well of a 96-well plate, 150 microliter of daily buffer (3 mg NADPH into 10 mL sodium phosphate buffer), 50microliter of DTNB solution, and 25 microliter of standards or samples will be added in quadruplicate, and the plate will be incubated at 37 °C for 3 minutes.Finally, 25 microliter GSSGR will be added to the previous mixture, and the plate will be read at 410 nm using a 96-well plate reader(UV spectrophotometer).

ELIGIBILITY:
Patients were included in the normal tension glaucoma group according to the following criteria.

Inclusion Criteria (normal tension glaucoma group):

* Clinical Diagnosis of Normal Tension Glaucoma: Patients underwent diurnal IOP phasing and were diagnosed as having normal tension glaucoma(IOP always lesser than 22 mm Hg by applanation tonometry), glaucomatous optic disc cupping on fundoscopic examination, open anterior chamber angles by gonioscopy(Schaffer grade III or more), and repeatable VF defects consistent with the diagnosis of glaucoma, according to results obtained with program 24-2 of the Humphrey Field Analyzer.
* Must be able to provide intravenous blood sampling

Exclusion Criteria (normal tension glaucoma group):

* Narrow iridocorneal angles
* Any evidence of secondary open-angle glaucoma
* Any other ocular disease except cataract
* History of previous intraocular surgery including cataract
* Any other systemic disease except hypertension

The control group was composed of age-matched healthy volunteers who had neither glaucoma nor other ocular diseases such as cataract, diabetic retinopathy or age related macular degeneration. The control group did not show any glaucomatous optic disc cupping on fundoscopic examination or visual field defects with program 24-2 of the Humphrey Field Analyzer. The healthy volunteers in the control group must be able to provide intravenous blood sampling.

Exclusion criteria for both groups:

* Smoking
* History of any chronic systemic disease with presumed low glutathione levels, including autoimmune diseases, alcoholic liver disease, cancer, and diabetes mellitus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of tertiary referred center
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Il Moon, Professor, Study Director — Department of Ophthalmology, St.Mary's Hospital, College of Medicine, The Catholic University of Korea
Locations (1):
- College of Medicine, The Catholic University of Korea, St. Mary's Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with normal tension glaucoma attending the glaucoma clinic of the Catholic Eye Center at the St. Mary' Hospital (Seoul, Korea) between June 2008 and October 2008, were recruited for this study. The control group was recruited from other age-gender-matched volunteers.
Pre-assignment Details: Only subjects who voluntarily wanted to participate in this study were recruited.
Groups:
- Normal Tension Glaucoma Group: Patients were diagnosed as having normal tension glaucoma if IOP measurements were lesser than 22 mm Hg by Goldmann applanation tonometry, characteristic glaucomatous cupping of the optic disc on fundoscopic examination, normal open anterior chamber angles by gonioscopy, and repeatable visual field defects consistent with the diagnosis of glaucoma, according to results obtained with program 24-2 of the Humphrey Field Analyzer (Carl Zeiss Meditec, Dublin, CA).
- Control Group: The control group was recruited from other age-gender-matched volunteers, and it was composed of subjects who had never neither glaucoma nor other ocular diseases such as cataract, diabetic ratinopathy, or age related macular degeneration.
Period: Overall Study
Arm/Group | Normal Tension Glaucoma Group | Control Group
Started | 19 | 30
Completed | 19 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Tension Glaucoma Group | Control Group | Total
Number analyzed (Participants) | 19 | 30 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 29 | 44
  >=65 years | 4 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 56.26 (8.48) | 52.70 (6.70) | 54.08 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 20 | 30
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 19 | 30 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Glutathione Levels
Description: Subjects were instructed to fast from midnight to 8 AM on the morning of the test. All blood samples were obtained by a qualified registered nurse in the morning, between 8 and 10 AM.
Time Frame: Once in the morning.
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Normal Tension Glaucoma Group | Control Group
Number analyzed (Participants) | 19 | 30
nmol | 524.02 (231.09) | 586.06 (156.08)

ADVERSE EVENTS:
Arm/Group | Normal Tension Glaucoma Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/30
Other Adverse Events (participants affected / at risk) | 0/19 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No